CLINICAL TRIAL: NCT04243733
Title: MTA vs CEM Pulpotomy in Young Permanent Molars With a Diagnosis of Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: MTA vs CEM Pulpotomy in Young Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Marwa Sharaan, Associate Professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110/2018
Record Dates: First submitted 2019-12-21; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — omega-Chloroacetophenone; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium enriched mixture material (CEM) (Other): Using CEM as a pulpotomy agent against MTA pulpotomy agent.
  Interventions: Other: CEM and MTA; Other: MTA and CEM
- Mineral trioxide aggregate material (MTA) (Experimental): Using MTA as a pulpotomy agent against CEM pulpotomy agent.
  Interventions: Other: CEM and MTA; Other: MTA and CEM

INTERVENTIONS:
Other: CEM and MTA — Pulpotomy agent
Other: MTA and CEM — Pulpotomy agent

SUMMARY:
The aim of the study

The purpose of this present clinical study will be to assess :

" the successful clinical outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis .

" the successful radiographic outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
Introduction and Review of Literature

Partial pulpotomy is generally regarded as the treatment of choice for immature teeth with exposed. pulp tissue. This treatment preserves pulp function,thus allowing continued root development . It was reported that 96% of teeth healed after being treated with partial pulpotomies associated with complicated crown fractures. This technique consists of the surgical amputation of 2-3mm of inﬂamed coronal pulp tissue. The wound surface is treated with a capping agent to promote healing and maintain viability of the remaining pulp tissue. It has been suggested that partial pulpotomy, compared with cervical pulpotomy, has many advantages including preservation of the cell-rich coronal pulp tissue, a necessary element for better healing , and the physiologic apposition of dentine in the coronal area. In contrast, cervical pulpotomy removes all the coronal pulp tissue, leaving the crown without the possibility of physiologic apposition of dentine, thereby increasing the risk of cervical fracture. Vital pulp treatment with materials such as mineral trioxide aggregate (MTA) are explored in studies on new trends in dental biomaterials .The successful use of MTA has been reported for partial pulpotomy of caries-exposed immature permanent teeth 5 and permanent teeth with irreversible pulpitits. On the other hand MTA possess some disadvantages; the most important one is its cost.

Calcium-enriched mixture (CEM, BioniqueDent, Tehran, Iran) cement has been introduced as a new endodontic biomaterial .This water-based tooth-colored cement is a biocompatible mixture cement that releases calcium and phosphate ions to form hydroxyapatite to induce the formation of a dentinal bridge.The product is alkaline (pH > 10.5) and releases calcium hydroxide during and after setting.The clinical use of CEM cement is similar to that of MTA. As a result, the characteristics of this cement are compared with MTA in some studies, showing a shorter setting and working time for CEM as well as a lower film thickness. CEM cement also shows a superior antibacterial effect 12 and improved handling 10. Both have similar sealing ability. The stated advantages of CEM cement and its potential effect on healing of the remaining pulp and the induction of dentinal bridge formation have led researchers to recommend use of the material in pulp treatment procedures in permanent teeth such as indirect and direct pulp cap, pulpotomy 13-17 and root-end fillings 18.One of the benefits of CEM cement is in the treatment of permanent teeth associated with irreversible pulpitis. The results of some clinical studies suggest vital pulp therapy with CEM as an alternative treatment to root canal therapy in such case with irreversible pulpitis.

To date, few studies have compared CEM cement and MTA as dressing materials for direct pulp cap and pulpotomy in young permanent molar teeth. The purpose of this present clinical study will be to assess the effect of CEM cement in the pulpotomy of young permanent molar teeth with irreversible pulpitis.

The aim of the study

The purpose of this present clinical study will be to assess :

" the successful clinical outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis .

" the successful radiographic outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis.

Materials and methods This is a double-blind, randomized, and con- trolled clinical trial. Forty children will be assigned randomly into two groups (20 children each) by block randomization, and allocation concealment will be done with closed envelop method. The sample size was obtained by using the G* power software statistical analysis according to previous studies. The research protocol will be approved by the Human Ethics Review Committee of the Faculty of Dentistry, Suez Canal University. For this 1-year clinical study, patients aged 6-14 years will be selected from the endodontic and pedodontic Clinics in the University. All of the parents will be told about the study and signed the informed consent.

Inclusion Criteria: Clinical examination reveals extended carious lesion on the molar teeth surface not extending toward the root. All of the patients report a history of pain typical of irreversible pulpitis ie; the chief complaints are of spontaneous pain lasting from a few seconds to several hours in the days before consultation. This radiating pain is exacerbated by hot and cold fluids and require analgesia for pain relief. The pain does not abate following tooth brushing or flossing. All of the parents are willing to join the study. All teeth are believed to be vital and the vitality of all the subjected molar teeth was checked by the operator during the pulpotomy procedure through visual inspection of pulpal hemorrhage.

Exclusion Criteria: Patients with systemic disease or physical or mental disability, extremely poor oral hygiene, periodontal problems, signs of abscess or fistula or non-physiological tooth mobility and non-restorable teeth will be excluded from the study. Teeth with external or internal root canal resorption, or root canal calcification in pre-treatment radiographs will be also excluded. Teeth where hemostasis can not be achieved will be excluded.

Pulpotomy Procedure: The treatment procedure will be performed after obtaining adequate local anesthesia with 2% lidocaine and 1/80,000 epinephrine ,the surface of the tooth was rinsed with normal saline and cleaned by swab wetted by a 0.2% chlorhexidine oral rinse . Pulpotomy procedures will be then performed with rubber dam then will be followed by complete removal of caries using fissure diamond burs and round stainless-steel burs. Pulpotomy will be performed with a sterile round diamond bur on a high-speed headpiece with copious water to remove all of the inflamed pulpal tissue. Following pulp amputation, the pulp chamber will be irrigated using 5% sodium hypochlorite until homeostasis is obtained. Teeth where hemostasis can not be achieved were excluded.

The CEM powder and liquid or MTA powder will be mixed according to the manufacturer's instruction and a base of approximately 2 mm of CEM cement will be placed over the amputation site. A wet cotton pellet will be used for adaption of the cement to the tooth walls. After 1 week the patient will be recalled for final restoration of the tooth with amalgam or a stainless steel crown. Prior to tooth restoration, the operator checks that the patient has no pain or clinical problems (ie; tenderness to percussion, swelling, fistula or mobility due to disease). A recall program is arranged for all patients and all of the teeth are evaluated clinically and radiographically.

Clinical Assessment: Clinical success is reviewed at 7 days and 3, 6 and 12 months after treatment. The teeth are tested for tenderness to percussion, soft tissue redness, dental swelling, abscess and fistula indicating any extension of inflammation toward the root canals. The parents are supplied with a telephone number so that they can inform the dentist of any problems.

Radiographic Assessment: No internal or external root resorption, no loss of lamina dura integrity, no periodontal ligament widening, and no alveolar bone resorption in the periapical region are considered indicative of successful treatment.

The clinical and radiographic assessments are all performed by the same two calibrated dentists. Where there initial is disagreement, consensus evaluations are performed by the two examiners.

ELIGIBILITY:
Inclusion Criteria:

- Clinical examination reveals extended carious lesion on the molar teeth surface not extending toward the root. All of the patients report a history of pain typical of irreversible pulpitis ie; the chief complaints are of spontaneous pain lasting from a few seconds to several hours in the days before consultation. This radiating pain is exacerbated by hot and cold fluids and require analgesia for pain relief. The pain does not abate following tooth brushing or flossing. All of the parents are willing to join the study. All teeth are believed to be vital and the vitality of all the subjected molar teeth was checked by the operator during the pulpotomy procedure through visual inspection of pulpal hemorrhage.

Exclusion Criteria:

* Clinical examination reveals extended carious lesion on the molar teeth surfaces not extending toward the root. All of the patients report a history of pain typical of irreversible pulpitis ie; the chief complaints are of spontaneous pain lasting from a few seconds to several hours in the days before consultation. This radiating pain is exacerbated by hot and cold fluids and require analgesia for pain relief. The pain does not abate following tooth brushing or flossing. All of the parents are willing to join the study. All teeth are believed to be vital and the vitality of all the subjected molar teeth was checked by the operator during the pulpotomy procedure through visual inspection of pulpal hemorrhage.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
the successful clinical outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis . | one year follow up after starting the case
  clinical signs and symptoms and testing sensibility of the pulp by cold test
the successful radiographic outcome of CEM cement in comparison to MTA in the pulpotomy of young permanent molar teeth with irreversible pulpitis. | one year follow up after starting the case
  healing of apical radiolucency, no occurrence of apical radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] References: [1] Smaïl-Faugeron V, Courson F, Durieux P, Muller-Bolla M, Glenny AM, Fron Chabouis H. Pulp treatment for extensive decay in primary teeth. Cochrane Database Syst Rev 2014; 8(8): CD003220. [2] Tannure PN, Azevedo CP, Barcelos R, Gleiser R, Primo LG. Long-term outcomes of primary tooth pulpectomy with and without smear layer removal: a randomized split-mouth clinical trial. Pediatr Dent 2011; 33(4): 316-20. [3] Barcelos R, Tannure PN, Gleiser R, Luiz RR, Primo LG. The influence of smear layer removal on primary tooth pulpectomy outcome: a 24-month, double-blind, randomized, and controlled clinical trial evaluation. Int J Paediatr Dent 2012; 22(5): 369-81. [4] McDougal RA, Delano EO, Caplan D, Sigurdsson A, Trope M. Success of an alternative for interim management of irreversible pulpitis. J Am Dent Assoc 2004; 135(12): 1707-12. [5] Barrieshi-Nusair KM, Qudeimat MA. A prospective clinical study of mineral trioxide aggregate for partial pulpotomy in cariously exposed permanent teeth. J Endod 2006; 32(8): 731-5. [6] Eghbal MJ, Asgary S, Baglue RA, Parirokh M, Ghoddusi J. MTA pulpotomy of human permanent molars with irreversible pulpitis. Aust Endod J 2009; 35(1): 4-8. [7] Holan G, Eidelman E, Fuks AB. Long-term evaluation of pulpotomy in primary molars using mineral trioxide aggregate or formocresol. Pediatr Dent 2005; 27(2): 129-36. [8] Noorollahian H. Comparison of mineral trioxide aggregate and formocresol as pulp medicaments for pulpotomies in primary molars. Br Dent J 2008; 204(11): E20. [9] Simancas-Pallares MA, Díaz-Caballero AJ, Luna-Ricardo LM. Mineral trioxide aggregate in primary teeth pulpotomy. A systematic literature review. Med Oral Patol Oral Cir Bucal 2010; 1(15): e 942-6. [10] Asgary S, Shahabi S, Jafarzadeh T, Amini S, Kheirieh S. The properties of a new endodontic material. J Endod 2008; 34(8): 990-3. [11] Amini Ghazvini S, Abdo Tabrizi M, Kobarfard F, Akbarzadeh Baghban A, Asgary S. Ion release and pH of a new endodontic cement, MTA and Portland cement. Iran Endod J 2009; 4(2): 74-8] [12] Asgary S, Kamrani FA. Antibacterial effects of five different root canal sealing materials. J Oral Sci 2008; 50(4): 469-74. [13] Asgary S, Eghbal MJ. Treatment outcomes of pulpotomy in permanent molars with irreversible pulpitis using biomaterials: a multi-center randomized controlled trial. Acta Odontol Scand 2013; 71(1): 130-6. [14] Asgary S, Eghbal MJ, Ghoddusi J, Yazdani S. One-year results of vital pulp therapy in permanent molars with irreversible pulpitis: an ongoing multicenter, randomized, non-inferiority clinical trial. Clin Oral Investig 2013; 17(2): 431-9. [15] Tabarsi B, Parirokh M, Eghbal MJ, Haghdoost AA, Torabzadeh H, Asgary S. A comparative study of dental pulp response to several pulpotomy agents. Int Endod J 2010; 43(7): 565-71. [16] Nosrat A, Asgary S. Apexogenesis of a symptomatic molar with calcium enriched mixture. Int Endod J 2010; 43(10): 940-4. [17] Nosrat A, Seifi A, Asgary S. Pulpotomy in caries-exposed immature permanent molars using calcium-enriched mixture cement or mineral trioxide aggregate: a randomized clinical trial. Int J Paediatr Dent 2013; 23(1): 56-63. [18] Asgary S, Eghbal MJ, Ehsani S. Periradicular regeneration after endodontic surgery with calcium-enriched mixture cement in dogs. J Endod 2010; 36(5): 837-41. [19] Asgary S, Eghbal MJ. The effect of pulpotomy using a calcium-enriched mixture cement versus one-visit root canal therapy on postoperative pain relief in irreversible pulpitis: a randomized clinical trial. Odontology 2010; 98(2): 126-33. [20] Faul, F., Erdfelder, E., Lang, A.-G., & Buchner, A. G*Power 3: A flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behavior Research Methods 2007; 39(2): 175-91.